CLINICAL TRIAL: NCT00132470
Title: AXIS IIa - Treatment With AX200 for Acute Ischemic Stroke
Brief Title: Treatment With AX200 for Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axaron Bioscience AG (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AX200_P2A_1
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke | interventions — Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: AX200 (G-CSF)

SUMMARY:
The AXIS study is a randomized, double-blind, placebo-controlled, dose-escalating phase IIa trial to investigate treatment with AX200 (granulocyte-colony stimulating factor; G-CSF) for acute ischemic stroke. The primary objective of the present phase IIa study is to assess the safety and tolerability of AX200 compared to placebo in subjects suffering from acute stroke. The secondary objective is to assess the effect of AX200 on subject outcome in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Stroke onset within 12 hours prior to start of study agent administration
* Ischemic stroke in the middle cerebral artery (MCA) territory confirmed by magnetic resonance imaging (MRI)

Exclusion Criteria:

* Time interval since stroke onset impossible to determine
* Carotid T-occlusion (magnetic resonance angiography [MRA])
* Subarachnoid hemorrhages
* Several safety parameters

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2004-12; Study Completion 2007-03

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Neurological outcome
ischemic lesion growth

CONTACTS AND LOCATIONS:
Overall Officials: Wolf-Rüdiger Schäbitz, MD, Principal Investigator — Universität Münster
Locations (2):
- Germany (2):
  - Neurology University of Heidelberg, Heidelberg
  - Neurology University of Muenster, Münster

REFERENCES:
- [Background] Schneider A, Kruger C, Steigleder T, Weber D, Pitzer C, Laage R, Aronowski J, Maurer MH, Gassler N, Mier W, Hasselblatt M, Kollmar R, Schwab S, Sommer C, Bach A, Kuhn HG, Schabitz WR. The hematopoietic factor G-CSF is a neuronal ligand that counteracts programmed cell death and drives neurogenesis. J Clin Invest. 2005 Aug;115(8):2083-98. doi: 10.1172/JCI23559. Epub 2005 Jul 7. PMID 16007267
- [Derived] Schabitz WR, Laage R, Vogt G, Koch W, Kollmar R, Schwab S, Schneider D, Hamann GF, Rosenkranz M, Veltkamp R, Fiebach JB, Hacke W, Grotta JC, Fisher M, Schneider A. AXIS: a trial of intravenous granulocyte colony-stimulating factor in acute ischemic stroke. Stroke. 2010 Nov;41(11):2545-51. doi: 10.1161/STROKEAHA.110.579508. Epub 2010 Oct 14. PMID 20947859